CLINICAL TRIAL: NCT02849769
Title: Medtronic Magnetic Resonance (MR) Conditional Tachyarrhythmia Therapy Products Post-approval Study
Brief Title: Magnetic Resonance (MR) Conditional Tachyarrhythmia Therapy Products Post-approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: MR Tachy PAS
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Tachyarrhythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients implanted with an MR-conditional Tachy device system: Patients implanted with an MR-conditional Tachy device system in the routine care
  Interventions: Device: Implant of an MR-conditional Tachy device system

INTERVENTIONS:
Device: Implant of an MR-conditional Tachy device system

SUMMARY:
Following product approval, further confirmation of the MR Conditional Tachyarrhythmia Therapy Systems sensing and detection performance post MRI exposure will be obtained by actively monitoring de-identified device data obtained through the Medtronic CareLink® Network.

DETAILED DESCRIPTION:
Pre-clinical testing and clinical data has demonstrated the safety and effectiveness of magnetic resonance (MR) Conditional Tachyarrhythmia Therapy Systems in the MR environment when used according to labeling requirements. Following approval, further confirmation of the MR Conditional Tachyarrhythmia Therapy Systems sensing and detection performance post MRI exposure will be obtained by actively monitoring de-identified device data obtained through the Medtronic CareLink® Network. MR conditional tachyarrhythmia therapy system enrolled in the Medtronic CareLink® Network (CL) will be used to prospectively assess spontaneous Ventricular Fibrillation (VF) episode detection following MRI exposure.

ELIGIBILITY:
Inclusion Criteria:

* MR conditional tachyarrhythmia therapy system enrolled in the Medtronic CareLink® Network (CL) will be used to prospectively assess spontaneous Ventricular Fibrillation (VF) episode detection following MRI exposure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MR conditional tachyarrhythmia therapy system enrolled in the Medtronic CareLink® Network (CL) will be used to prospectively assess spontaneous Ventricular Fibrillation (VF) episode detection following MRI exposure.
Sampling Method: Non-Probability Sample
Enrollment: 10979 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The proportion of episodes with ≥ 5 seconds VF detection delay in the MR conditional tachyarrhythmia therapy system following MRI exposure. | up to 5 years post-approval.
  The primary objective will be analyzed and reported when 50 patients with a true VF episode following MR exposure have been identified

SECONDARY OUTCOMES:
The number of patients with 2 or more scans | up to 5 years post-approval
  The estimate of patients receiving multiple MRI scans will include all patients regardless if the patient has experienced a VF episode.
Pre-MRI and post-MRI LV lead PCT measurements obtained through CareLink | up to 5 years post-approval
  Pre-MRI and post-MRI LV lead PCT measurements obtained through CareLink will be summarized for MR CRT-D patients. Summary statistics will be presented separately for pre-MRI and post-MRI PCT measurements

CONTACTS AND LOCATIONS:
Overall Officials: Product Surveillance Registry Medtronic Product Surveillance Registry, Study Chair — Medtronic